CLINICAL TRIAL: NCT03592277
Title: Vitamins B1 and C to Improve Outcomes in Patients With Severe Sepsis
Brief Title: Vitamin C & Thiamine to Treat Sepsis and Septic Shock
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SF-18-42
Record Dates: First submitted 2018-06-18; First posted 2018-07-19 (Actual); Results first posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Sepsis; Septic Shock
Keywords: Sepsis; Septic Shock; Vitamin C; Thiamine
MeSH Terms: conditions — Sepsis; Shock, Septic | interventions — Ascorbic Acid; Thiamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All parties involved, except for pharmacy personnel will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TREATMENT with Vitamins C and B1 (Experimental): Patients in the Vitamins C and B1 arm will receive 1.5g of vitamin C in 100mL of 0.9% sodium chloride (normal saline) every six hours for four days or until discharge from the ICU, whichever happens first (seventeen dose maximum). In addition, they will receive 200 mg IV vitamin B1 every 12 hours in 50 mL of normal saline for four days or until ICU discharge (whichever happens first, nine dose maximum).
  Interventions: Drug: Vitamin C; Drug: Vitamin B1
- PLACEBO with saline only (No Intervention): Patients in the placebo (control group) arm will receive the 100 mL of 0.9% sodium chloride every six hours and 50 mL of 0.9% sodium chloride every 12 hours to act as placebos for the vitamins C and B1 respectively.

INTERVENTIONS:
Drug: Vitamin C — Patients will receive 1.5g of vitamin C in 100mL of 0.9% sodium chloride (normal saline) every six hours for four days or until discharge from the ICU, whichever happens first (seventeen dose maximum).
  Other Names: Ascorbic Acid
  Arms: TREATMENT with Vitamins C and B1
Drug: Vitamin B1 — Patients will also receive 200 mg of IV vitamin B1 every 12 hours in 50 mL of normal saline for four days or until ICU discharge (whichever happens first, nine dose maximum).
  Other Names: Thiamine
  Arms: TREATMENT with Vitamins C and B1

SUMMARY:
Investigators propose to investigate the use of IV vitamins B1 and C in a randomized, double-blinded, prospective trial to determine if these medications decrease mortality rates in patients with severe sepsis or septic shock.

DETAILED DESCRIPTION:
Investigators propose to investigate the use of IV vitamins B1 and C in a randomized, double-blinded, prospective trial to determine if these medications decrease mortality rates in patients with severe sepsis or septic shock. Patients experiencing evidence-based diagnoses of sepsis and severe sepsis and septic shock will be randomized to the two study arms for care, and all other care left to decisions of intensive care teams.

ELIGIBILITY:
Patients must meet all inclusion criteria:

1. Between the ages of 18 and 90 years old
2. Have severe sepsis or septic shock. Severe sepsis and septic shock will be defined by the Surviving Sepsis 2012 guidelines.
3. Weight more than 30 kg
4. Full code

Exclusion Criteria:

1. Not diagnosed with severe sepsis or septic shock
2. Younger than 18 or older than 90 years old
3. With a history of nephrolithiasis
4. Who are pregnant
5. Weigh less than 30 kg
6. Not located in the ICU
7. Do not resuscitate (DNR) or do not intubate (DNI), no escalation of care, or comfort measures only (CMO)
8. Currently on dialysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2021-02-22 (Actual); Study Completion 2021-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Shapiro, MD, Principal Investigator — Saint Francis Hospital and Medical Center
Locations (1):
- Saint Francis Hospital and Medical Center, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients admitted to the intensive care unit with a diagnosis of septic shock were identified by study team members, offered for recruitment, recruited and randomized upon arrival to the unit. This began September 14, 2018 and the final recruitment occurred on February 22, 2021.
Pre-assignment Details: The only exclusions for for patients who opted out of the study following initial consent. No other run-in events occurred.
Groups:
- Vitamins C and B1: Patients in this arm will receive 1.5g of vitamin C in 100mL of 0.9% sodium chloride (normal saline) every six hours for four days or until discharge from the ICU, whichever happens first (seventeen dose maximum). In addition, they will receive 200 mg IV vitamin B1 every 12 hours in 50 mL of normal saline for four days or until ICU discharge (whichever happens first, nine dose maximum).
  Vitamin C: Patients will receive 1.5g of vitamin C in 100mL of 0.9% sodium chloride (normal saline) every six hours for four days or until discharge from the ICU, whichever happens first (seventeen dose maximum).
  Vitamin B1: Patients will also receive 200 mg of IV vitamin B1 every 12 hours in 50 mL of normal saline for four days or until ICU discharge (whichever happens first, nine dose maximum).
- Placebo: Patients in the control arm will receive the 100 mL of 0.9% sodium chloride every six hours and 50 mL of 0.9% sodium chloride every 12 hours to act as placebos for the vitamins C and B1 respectively.
Period: Overall Study
Arm/Group | Vitamins C and B1 | Placebo
Started | 60 | 60
Powered For | 60 | 60
Completed | 54 | 52
Not Completed | 6 | 8
Not completed — Withdrawal by Subject | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamins C and B1 | Placebo | Total
Number analyzed (Participants) | 54 | 52 | 106
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 22 | 47
  >=65 years | 29 | 30 | 59
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58 to 74] | 69 [54.5 to 78] | 67 [57 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 23 | 51
  Male | 26 | 29 | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 54 | 52 | 106
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (7.6) | 29.7 (7.6) | 29.0 (7.6)

OUTCOME MEASURES:

1. Primary Outcome: Mortality Rates
Description: All-cause mortality from time of enrollment/treatment to 30 days post hospital discharge (up to 87 days)
Time Frame: From time of treatment to 30 days post hospital discharge, up to 87 days.
Measure: Count of Participants; unit: Participants
Groups:
- Vitamins C and B1: Patients in this arm will receive 1.5g of vitamin C in 100mL of 0.9% sodium chloride (normal saline) every six hours for four days or until discharge from the ICU, whichever happens first (seventeen dose maximum). In addition, they will receive 200 mg IV vitamin B1 every 12 hours in 50 mL of normal saline for four days or until ICU discharge (whichever happens first, nine dose maximum).
  Patients may remain in the ICU and/or hospitalized after completing 4 days of treatment.
  Vitamin C: Patients will receive 1.5g of vitamin C in 100mL of 0.9% sodium chloride (normal saline) every six hours for four days or until discharge from the ICU, whichever happens first (seventeen dose maximum).
  Vitamin B1: Patients will also receive 200 mg of IV vitamin B1 every 12 hours in 50 mL of normal saline for four days or until ICU discharge (whichever happens first, nine dose maximum).
Arm/Group | Vitamins C and B1 | Placebo
Number analyzed (Participants) | 54 | 52
Participants | 12 | 7
Statistical Analysis 1: Comparison: Vitamins C and B1 vs Placebo; Test type: Superiority; p = 0.344, Chi-squared

2. Secondary Outcome: Hospital Length of Stay
Description: Total number of days patient is admitted to the hospital
Time Frame: From admission to the hospital through hospital discharge, up to 57 days.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Vitamins C and B1 | Placebo
Number analyzed (Participants) | 54 | 52
days | 8.5 [7.0 to 13.0] | 7.0 [5.5 to 11.5]
Statistical Analysis 1: Comparison: Vitamins C and B1 vs Placebo; Test type: Superiority; p = 0.526, Chi-squared

3. Secondary Outcome: Intensive Care Unit Length of Stay
Description: Total number of days patient is admitted to the ICU
Time Frame: From time of admission to the ICU through discharge from the ICU, up to 25 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Vitamins C and B1 | Placebo
Number analyzed (Participants) | 54 | 52
days | 3.5 [2.0 to 7.0] | 3.0 [2.0 to 4.0]
Statistical Analysis 1: Comparison: Vitamins C and B1 vs Placebo; Test type: Superiority; p = 0.123, Chi-squared

4. Secondary Outcome: Readmission Rate
Description: Readmission to the hospital within 30 days after discharge
Time Frame: 30 days after hospital discharge
Population: 54 patients received treatment, 11 died during initial admission and therefore excluded from readmission statistics. Of the 52 patients in the control group 7 died during initial admission and were excluded from readmission statistics. One control patient was withdrawn and also could not be considered for readmission statistics.
Measure: Number; unit: participants
Arm/Group | Vitamins C and B1 | Placebo
Number analyzed (Participants) | 43 | 44
participants | 17 | 15
Statistical Analysis 1: Comparison: Vitamins C and B1 vs Placebo; Test type: Superiority; p = 0.660, Fisher Exact

5. Secondary Outcome: Ventilator Days
Description: Number of days patient required ventilator
Time Frame: From admission to the ICU through discharge from the ICU, up to 25 days.
Population: Intervention arm-1 patient made CMO and terminally extubated, 1 patient had insufficient data. Control-3 patients made CMO then terminally extubated
Measure: Mean (Standard Deviation); unit: days on ventilator
Arm/Group | Vitamins C and B1 | Placebo
Number analyzed (Participants) | 52 | 49
days on ventilator | 2.6 (3.5) | 2.3 (5.8)
Statistical Analysis 1: Comparison: Vitamins C and B1 vs Placebo; Test type: Superiority; p = 0.745, t-test, 2 sided

6. Secondary Outcome: Hours on Vasopressors
Description: Number of hours patient required vasopressors in norepinephrine equivalence.
Time Frame: From admission to the ICU through discharge from the ICU, up to 25 days.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Vitamins C and B1 | Placebo
Number analyzed (Participants) | 54 | 52
Hours | 50.0 (9.8) | 35.9 (6.5)
Statistical Analysis 1: Comparison: Vitamins C and B1 vs Placebo; Test type: Superiority; p = 0.236, Chi-squared

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of enrollment into the study, during hospital stay and continued until 30 days following discharge from the hospital, up to 87 days.
Arm/Group | Vitamins C and B1 | Placebo
All-Cause Mortality (participants affected / at risk) | 12/54 | 7/52
Serious Adverse Events (participants affected / at risk) | 17/54 | 15/52
Other Adverse Events (participants affected / at risk) | 0/54 | 0/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamins C and B1 (N=54) | Placebo (N=52)
Death due to sepsis or septic shock (Infections and infestations) | 12 (12) | 7 (7)
Readmissions within 30 days (Infections and infestations) | 17 (17) | 15 (15) — Readmissions within 30 days of index hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/77/NCT03592277/Prot_SAP_000.pdf